CLINICAL TRIAL: NCT02744079
Title: A Pilot Presurgical Trial of Insulin Inhibition by a Ketogenic Diet in Operable Breast Cancer
Brief Title: Comparison of Healthy Diets on Breast Cancer Markers
Acronym: KetoBreast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Eugene Fine, Professor of Radiology, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-6346
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Breast Neoplasms
Keywords: diet; dietary intervention; carbohydrate restriction; low carbohydrate; fat restriction; low fat; cancer; breast cancer; pre-surgical window; biomarker
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low carbohydrate diet (Active Comparator): 45 subjects will receive a very low carbohydrate diet between a positive breast biopsy and surgical tumor removal
  Interventions: Behavioral: Low carbohydrate diet
- Low fat diet (Active Comparator): 20 subjects will receive a lo fat diet between a positive breast biopsy and surgical tumor removal
  Interventions: Behavioral: Low fat diet

INTERVENTIONS:
Behavioral: Low carbohydrate diet — 45 subjects will be randomized to a dietary arm consisting of a complete, prepared very low carbohydrate diet, delivered to their homes, for the interval between positive breast biopsy and surgical tumor removal
  Arms: Low carbohydrate diet
Behavioral: Low fat diet — 20 subjects will be randomized to a dietary arm consisting of a complete, prepared low fat diet, delivered to their homes, for the interval between positive breast biopsy and surgical tumor removal.
  Arms: Low fat diet

SUMMARY:
Women post breast mass biopsy with ER+or ER- cancer will be randomized to two diets--goal of 45 of them to a ketogenic insulin inhibiting diet, 20 to a low fat diet with whole grains and fruits and vegetables. The initial biopsy will be evaluated along with the surgical specimen pathology to compare changes in biomarkers, particularly of proliferation (Ki-67) and apoptosis (TUNEL).

DETAILED DESCRIPTION:
A healthy diet has been defined in various ways. The investigators wish to compare the effects of two diets on ER positive breast cancer tissues. The diets will be administered between the time of diagnosis and the time of surgical removal. Both diets have been proposed as healthy, but differ in their composition. One constitutes a low fat diet with extra fiber, fruits and vegetable servings, while the other comprises a diet low in carbohydrate content, aiming to lower insulin secretion. Patients will be randomized to each group, with 20 assigned to the low fat arm and 45 to the low carbohydrate arm.

ELIGIBILITY:
Inclusion Criteria:

Women with biopsy proven breast cancer.

Exclusion Criteria:

-

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
TUNEL comparison of each dietary intervention at surgical removal to measure change in apoptosis in tumor cells | 2 years
Ki-67 comparison of each dietary intervention at surgical removal to measure change in proliferation of tumor cells | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eugene J Fine, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- The Albert Einstein College of Medicine of Yeshiva University, The Bronx, New York, United States

REFERENCES:
- [Background] Fine EJ, Segal-Isaacson CJ, Feinman RD, Herszkopf S, Romano MC, Tomuta N, Bontempo AF, Negassa A, Sparano JA. Targeting insulin inhibition as a metabolic therapy in advanced cancer: a pilot safety and feasibility dietary trial in 10 patients. Nutrition. 2012 Oct;28(10):1028-35. doi: 10.1016/j.nut.2012.05.001. Epub 2012 Jul 26. PMID 22840388
- [Background] Jain R, Strickler HD, Fine E, Sparano JA. Clinical studies examining the impact of obesity on breast cancer risk and prognosis. J Mammary Gland Biol Neoplasia. 2013 Dec;18(3-4):257-66. doi: 10.1007/s10911-013-9307-3. Epub 2013 Nov 13. PMID 24221746
- [Background] Fine EJ, Miller A, Quadros EV, Sequeira JM, Feinman RD. Acetoacetate reduces growth and ATP concentration in cancer cell lines which over-express uncoupling protein 2. Cancer Cell Int. 2009 May 29;9:14. doi: 10.1186/1475-2867-9-14. PMID 19480693